CLINICAL TRIAL: NCT05640739
Title: The Effect of Demonstration and Video Viewing Education on Metered Dose Inhaler Usage Skills in Asthma Patients: A Randomized Controlled Study
Brief Title: The Effect of Demonstration and Video Viewing Education on Metered Dose Inhaler Usage Skills in Asthma Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The work could not be completed due to the earthquake in Kahramanmaraş.
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Yasemin SAZAK, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HasanKU-SAZAK-002
Record Dates: First submitted 2022-11-27; First posted 2022-12-07 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Asthma; Patient Education
Keywords: Metered Dose Inhalers; Patient Education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group patients (No Intervention): Data will be collected from the patients in the control group without any application and their ability to use MDI will be evaluated.
- Demonstration group patients (Experimental): Patients in the demonstration group will be given inhaler training (practically) by the researcher. The training will include steps compatible with the video. After the training, the patients will be asked to use inhaler drugs again, and their skill scores will be re-evaluated and the mistakes made by the patients will be shown by the researcher in the demonstration group. On the 7th day of the study, the patients will be called by the researcher with a video call, and the patients will be asked to use their MDI drugs again, and the MDI use skill chart will be filled again.
  Interventions: Behavioral: Demonstration method for the use of the Metered Dose Inhaler
- Video group patients (Experimental): The patients in the video group will be shown the video of using MDI prepared by the researchers. The training will be completed by watching the MDI usage video prepared by the researchers in the patients in the video group. After the training, the patients will be asked to use the inhaler again and their skill scores will be re-evaluated. Their mistakes will be shown by making them watch it again from the video. On the 7th day of the study, the patients will be called by the researcher with a video call, and the patients will be asked to use their MDI drugs again, and the MDI use skill chart will be filled again.
  Interventions: Behavioral: Video watching method for the use of the Metered Dose Inhaler

INTERVENTIONS:
Behavioral: Demonstration method for the use of the Metered Dose Inhaler — The effectiveness of the training given by the demonstration method for the use of the Metered Dose Inhaler (MDI)
  Arms: Demonstration group patients
Behavioral: Video watching method for the use of the Metered Dose Inhaler — The effectiveness of the training given by video watching method for the use of the Metered Dose Inhaler (MDI)
  Arms: Video group patients

SUMMARY:
In the treatment of respiratory diseases such as COPD and asthma, bronchodilators and steroids, which are essential drugs, are preferred to be administered by inhalation compared to oral and parenteral routes. In the studies conducted with the use of inhaler drugs, it is seen that many wrong practices have been made regarding the techniques of using the inhaler drugs and that the correct usage techniques are not followed. Inability to use the inhaler device fully and correctly; It causes consequences such as failure to control the disease, increase in drug use and side effects, increase in exacerbations, high hospitalization and waste of drugs, both undermining the trust in treatment and putting an extra burden on the health expenditures of the countries. This research aim is to evaluate the effectiveness of the training given with the demonstration method and video watching method for the use of the Metered Dose Inhaler (MDI) in asthmatic patients, and to ensure that the patients learn the correct inhaler use techniques.

DETAILED DESCRIPTION:
The research was planned as a randomized controlled experimental study. Patients who applied to the Elbistan State Hospital chest polyclinic with a diagnosis of asthma and met the criteria for inclusion in the study will be divided into control group, demonstration training group and video surveillance training groups. Simple randomization method will be used to determine the groups. The sample of the research; With G-Power, it was determined as 21 people for each group at 80% power, 5% error and 95% confidence interval. To prevent data loss; It was decided to have 32 people in the control group, 32 people in the demonstration training group, and 32 people in the video watching training group. After informing the patients about the study, the consent of the patients who agreed to participate in the study will be obtained and the research data will be collected by face-to-face interview method. After the patient identification form is completed, the patients will be asked to use the MDI inhaler and the MDI use skills chart will be filled. For the steps of MDI use, it will be evaluated with the use of MDI skill chart based on the Thoracic Society National Asthma Diagnosis and Treatment Guidelines. The total skill scores will be determined by giving 1 point for the correct application and 0 points for the incorrect application. Data will be collected from the patients in the control group without any application and their ability to use MDI will be evaluated. Patients in the demonstration group will be given inhaler training (practically) by the researcher. The training will include steps compatible with the video. The training will be completed by watching the MDI usage video prepared by the researchers in the patients in the video group. After the training, the patients will be asked to use the inhaler again, and their skill scores will be re-evaluated, and the mistakes made by the patients will be shown by the researcher in the demonstration group, and in the video group by allowing them to watch the video again. The patients in the control group will fill out the MDI skill form again (after 30 minutes) without any procedure. To prevent drug overdose, patients will be administered with placebo training drugs. The patients in the whole group will be called by the researcher on the 7th day of the study, and the patients will be asked to use their MDI drugs again, and the MDI use skill chart will be filled again. The control group will then be given inhaler training by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed asthma diagnosis
* be 18 years or older,
* Using MDI,
* Volunteer to participate in the research.
* Patients who do not have communication problems,
* Patients who can make video calls,

Exclusion Criteria:

* Not complying with the principle of volunteering
* Answering data collection forms incompletely
* Patients who did not answer calls for the last test and could not be reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-12 (Estimated); Primary Completion 2023-03-12 (Estimated); Study Completion 2023-05-12 (Estimated)

PRIMARY OUTCOMES:
MDI Use Skills Chart | Baseline (Before training)
  For the steps of MDI use, it will be evaluated with the use of MDI skill chart based on the Thoracic Society National Asthma Diagnosis and Treatment Guidelines. The total skill scores will be determined by giving 1 point for the correct application and 0 points for the incorrect application.
MDI Use Skills Chart | Immediately after training
  For the steps of MDI use, it will be evaluated with the use of MDI skill chart based on the Thoracic Society National Asthma Diagnosis and Treatment Guidelines. The total skill scores will be determined by giving 1 point for the correct application and 0 points for the incorrect application.
MDI Use Skills Chart | 7th day after training
  For the steps of MDI use, it will be evaluated with the use of MDI skill chart based on the Thoracic Society National Asthma Diagnosis and Treatment Guidelines. The total skill scores will be determined by giving 1 point for the correct application and 0 points for the incorrect application.

CONTACTS AND LOCATIONS:
Overall Officials: Nermin OLGUN, Professor, Principal Investigator — Hasan Kalyoncu University Faculty of Nursing; Keriman AYTEKIN KANADLI, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No